CLINICAL TRIAL: NCT07316920
Title: An Exploratory Clinical Study of the Safety and Efficacy of RN1701 Injection in the Treatment of Relapsed/Refractory B-Cell Lymphomas
Brief Title: A Clinical Study of of RN1701 Injection in the Treatment of Relapsed/Refractory B-Cell Lymphomas
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: YANRU WANG (Other)
Collaborators: Allorunning Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, YANRU WANG, Clinical Professor, Affiliated Hospital of Jiangsu University
Organization: Affiliated Hospital of Jiangsu University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN1701JB
Record Dates: First submitted 2025-12-09; First posted 2026-01-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory B-cell Lymphoma
Keywords: Relapsed/refractory; B-cell lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed/refractory B-cell lymphoma (Experimental): Relapsed/refractory B-cell lymphoma patients to be treated with RN1701 cells.
  Interventions: Biological: RN1701 injection

INTERVENTIONS:
Biological: RN1701 injection — RN1701 injection is a bispecific CD19/CD20-targeted allogeneic CAR-T. A single infusion of CAR-T cells will be administered intravenously

SUMMARY:
This single-arm, open-label pilot study will assess the safety and efficacy of RN1701, a bispecific CD19/CD20-targeted allogeneic CAR-T-cell product, in patients with relapsed or refractory B-cell lymphoma. Up to 19 participants will be enrolled in a conventional 3 + 3 dose-escalation scheme. The primary objective of the study is to evaluate the safety and feasibility of RN1701 for the treatment of relapsed/refractory B-cell lymphoma. The secondary objective is to evaluate the efficacy of RN1701 for the treatment of relapsed/refractory B-cell lymphoma. The exploratory objective is to evaluate the expansion, persistence, and ability of RN1701 to deplete CD19- and/or CD20-positive cells in patients with relapsed/refractory B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation; full understanding of the study and provision of written informed consent obtained before any study-related procedure not part of standard care; willingness to comply with follow-up.
2. Age 18-75 years; either sex.
3. ECOG performance status 0-1.
4. Histologically confirmed large B-cell lymphoma, follicular lymphoma, mantle-cell lymphoma, or indolent lymphoma transformed to DLBCL; CD19 and/or CD20 positive.
5. At least one measurable lesion per Lugano criteria: nodal lesion longest diameter >1.5 cm, extranodal lesion >1.0 cm.
6. Prior treatment response must meet one of the following:

   • Large B-cell lymphoma, grade 3B follicular lymphoma, transformed indolent lymphoma: i. Primary refractory and ineligible/unable to receive autologous CAR-T: best response PD after ≥2 cycles of first-line therapy, or SD after ≥4 cycles.

   ii. Relapse ≤12 months after achieving CR with first-line chemo-immunotherapy. iii. Relapse/progression ≤12 months after autologous HSCT. iv. Refractory to, relapsed after, or progressed on ≥2 prior lines (including autologous CAR-T): best response PD or SD after ≥2 cycles of the most recent regimen.

   v. Transformed indolent lymphoma: prior chemotherapy for iNHL and ≥1 systemic regimen after transformation, fulfilling the above refractory/relapse criteria.

   • Grade 1, 2, or 3A follicular lymphoma: i. Primary refractory and ineligible/unable to receive autologous CAR-T: best response PD after ≥2 cycles of first-line therapy.

   ii. Refractory to, relapsed after, or progressed on ≥2 prior lines (including autologous CAR-T): best response PD or SD after ≥2 cycles of the most recent regimen.

   • Mantle-cell lymphoma: i. Primary refractory and ineligible/unable to receive autologous CAR-T: best response PD after ≥2 cycles of first-line therapy, or SD after ≥4 cycles.

   ii. Refractory to, relapsed after, or progressed on ≥2 prior lines (including autologous CAR-T): best response PD or SD after ≥2 cycles of the most recent regimen.
7. Estimated life expectancy ≥3 months.
8. Screening laboratory values (may be repeated once):

   * Hemoglobin ≥8.0 g/dL (no transfusion within 7 days).
   * Platelets ≥50×10⁹/L (no transfusion within 7 days).
   * ANC ≥1.0×10⁹/L (growth-factor support allowed if none within 7 days of test).
   * AST/ALT ≤3×ULN (≤5×ULN if liver involvement).
   * Serum creatinine ≤1.5×ULN or CrCl ≥60 mL/min (Cockcroft-Gault).
   * Total bilirubin ≤2×ULN (≤3×ULN if liver involvement); except congenital bilirubin disorders (e.g., Gilbert's syndrome: direct bilirubin ≤1.5×ULN).
   * INR, PT, APTT <1.5×ULN.
9. Toxicities from prior anti-cancer therapy (except alopecia, nausea, and the above lab values) must have stabilized at baseline or resolved to ≤Grade 1.
10. WOCBP must have a negative high-sensitivity serum β-hCG pregnancy test at screening and again before the first dose of cyclophosphamide/fludarabine.
11. Subjects of reproductive potential must use effective contraception for ≥12 months after completing study therapy.

Exclusion Criteria:

* Subjects with any of the following conditions are ineligible for this trial:

  1. Any malignancy other than B-cell non-Hodgkin lymphoma ever diagnosed or treated, except:

     * Malignancy that received curative therapy and has shown no evidence of active disease for ≥2 years before enrolment; or
     * Adequately treated non-melanoma skin cancer with no current evidence of disease.
  2. Prior anti-cancer therapy within the stated windows (before lymphodepletion):

     * CNS prophylaxis (e.g., intrathecal methotrexate and/or cytarabine) within 7 days;
     * Cytotoxic chemotherapy or radiotherapy within 14 days;
     * Small-molecule targeted or epigenetic therapy within 14 days or 5 half-lives, whichever is longer;
     * Monoclonal antibody, bispecific antibody, or antibody-drug conjugate within 21 days or 5 half-lives, whichever is shorter;
     * Investigational drug or invasive investigational device within 28 days (if the therapy is also investigational, the 28-day wash-out applies);
     * Autologous haematopoietic stem-cell transplant or CD19-directed autologous CAR-T therapy within 100 days.
  3. Any autologous cellular or gene therapy other than CD19-directed autologous CAR-T.
  4. Any allogeneic cellular (including CAR-T) or gene therapy.
  5. Prior allogeneic haematopoietic stem-cell transplantation.
  6. Positive donor-specific antibody (DSA).
  7. At least one of the following high-risk features:

     * Sum of the product of perpendicular diameters (SPD) of all measurable lesions ≥100 cm²;
     * Bulky disease: single mass ≥7.5 cm; mediastinal mass with maximum diameter >1/3 of thoracic diameter;
     * Obstructive/compressive emergency (e.g., bowel obstruction, vascular compression) requiring urgent intervention at screening.
  8. Active CNS involvement (symptomatic or positive CSF/imaging); subjects with prior CNS disease now in remission (asymptomatic with negative CSF and imaging) are eligible.
  9. Significant bleeding diathesis: gastrointestinal bleeding, haemorrhagic cystitis, coagulopathy, hypersplenism (splenomegaly on exam/US, cytopenias, hyperplastic marrow) or ongoing anticoagulation.
  10. Chronic concomitant systemic corticosteroids or other immunosuppressants, except: topical, ocular, intra-articular, nasal or inhaled corticosteroids; short-course steroids for prophylaxis (e.g., contrast allergy).
  11. Severe underlying medical conditions:

      * Active serious viral, bacterial or uncontrolled systemic fungal infection;
      * Active systemic autoimmune disease requiring therapy.
  12. Significant cardiac disease:

      * NYHA class III or IV congestive heart failure;
      * Myocardial infarction or CABG within 6 months before enrolment;
      * Clinically relevant ventricular arrhythmia or unexplained syncope not vasovagal or dehydration-related;
      * Severe non-ischaemic cardiomyopathy;
      * Left ventricular ejection fraction (LVEF) <45% by echo or MUGA within 4 weeks before lymphodepletion.
  13. Resting oxygen saturation <92%.
  14. Clinically relevant prior or current CNS disorder: epilepsy, seizure-like episodes, paralysis, aphasia, stroke, severe head trauma, dementia, Parkinson's disease, cerebellar disorder, organic brain syndrome or major psychiatric illness.
  15. Live-attenuated vaccine within 4 weeks before screening.
  16. Major surgery within 2 weeks before screening or planned within 2 weeks after study treatment (local anaesthesia allowed).
  17. Positive screen for HBsAg, HBeAg, HBV DNA, HCV antibody, HCV RNA, or HIV antibody.
  18. Life-threatening allergy, hypersensitivity or intolerance to study-drug excipients including, but not limited to, DMSO.
  19. Lactating women.
  20. Any condition that, in the investigator's opinion, renders the subject unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Toxicity and adverse-event grading after RN1701 treatment | up to 12 months after infusion
  all toxicities and AEs will be assessed according to the National Cancer Institute CTCAE v5.0
CRS grading after RN1701 treatment | up to 12 months after infusion
  Cytokine Release Syndrome (CRS) will be graded using the Lee DW et al. CRS grading scale.
  Grade 1: Fever, mild symptoms, manageable with supportive care Grade 2: Moderate symptoms (eg, hypotension, hypoxia), requires intervention (eg, intravenous fluids, antipyretics) Grade 3: Severe symptoms (eg, multiorgan involvement), requires corticosteroids and tocilizumab Grade 4: Life-threatening, requires intensive care unit (ICU) care and urgent interventions

SECONDARY OUTCOMES:
Overall response rate (ORR = CR + PR) of patients receive RN1701 treatment | 1, 3, 6, and 12 months after infusion
  according to the Lugano criteria and CSCO guidelines
Disease control rate (DCR = CR + PR + SD) of patients receive RN1701 treatment | 1, 3, 6, and 12 months after infusion
  according to the Lugano criteria and CSCO guidelines
Assessment includes contrast-enhanced CT of head/neck, chest, abdomen, and pelvis, plus whole-body PET-CT | 1, 3, 6, and 12 months after infusion
  Tumor measurements and evaluations must be performed with the same technique used at baseline
CAR copies and cell count of CAR-T in blood after RN1701 treatment | Days 0, 1, 3, 5, 7, 9, 11, 14, 21, 28 and month 2, 3, 6, 9, 12 after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No